CLINICAL TRIAL: NCT06292468
Title: Effects of Plantar Cutaneous Sensory Stimulation on Foot Tactile Sensitivity, Postural Control, and Spatiotemporal Gait Parameters in Patients With Diabetic Neuropathy
Brief Title: Plantar Cutaneous Sensory Stimulation in Patients With Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0238
Record Dates: First submitted 2024-01-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetic neuropathy; Gait parameters; Plantar cutaneous stimulation; Postural instability
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy (Active Comparator): This group received conventional physical therapy protocol along with foot care guidelines.
  Interventions: Other: Traditional physical therapy
- Plantar cutaneous sensory stimulation. (Experimental): This group received plantar cutaneous sensory stimulation along with conventional physical therapy protocol and foot care guidelines.
  Interventions: Other: Plantar cutaneous sensory stimulation

INTERVENTIONS:
Other: Traditional physical therapy — This group received 30 minutes of muscle stretching (quadriceps, gastrocnemius, hamstrings, tibialis), bilateral ankle strengthening, gait training and foot care guidelines, 3 times a week for a duration of six weeks.
  Arms: Traditional physical therapy
Other: Plantar cutaneous sensory stimulation — This group received 45 minutes of plantar cutaneous sensory stimulation, TENS, muscle stretching (quadriceps, gastrocnemius, hamstrings, tibialis), bilateral ankle strengthening, gait training, and foot care guidelines, 3 times a week for a duration of six weeks.
  Arms: Plantar cutaneous sensory stimulation.

SUMMARY:
To determine the effects of plantar cutaneous sensory stimulation on foot tactile sensitivity, postural control, and spatiotemporal gait parameters in patients with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged between 45-67 years.
* Both male and female genders are included.
* DM for the past 7 years.
* Scored > 2/13 on the Michigan Neuropathy Screening Instrument (MNSI) questionnaire including at least two DPN symptoms.
* Scored >1/10 on MNSI physical assessment including impaired vibration perception

Exclusion Criteria:

* Loss of protective foot sensation (defined as a lack of response to the monofilament of the sensory evaluation instrument).
* Comorbidities include visual impairment, cerebrovascular accident, orthopedic trauma, labyrinthitis, peripheral vascular disease, and heart failure.
* Foot ulcers, orthopedic or surgical problems in a lower limb, other neurological impairment.
* Use of assistive devices for ambulation.
* Inability to walk independently with or without an assistive device.
* Receiving any structured supervised physiotherapy intervention

Ages: 45 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Foot tactile sensitivity | 6th week
  Semmes Weinstein monofilaments, Foot tactile sensitivity loss, commonly assessed by monofilaments, is a fall risk factor among older adults. The broadly used threshold of the monofilament for fall risk assessment in older adults is 5.07
Postural control | 6th week
  Brief BESTest is a clinical balance assessment tool. It is an abbreviated version of Balance Evaluation Systems Test (BESTest) designed to assess 6 different aspects contributing to postural control in standing and walking. It consist of 27 tasks, with 36 items in total. Each items is scored based on ordinal scale scoring from 0- 3 where 3 representing best performances and 0 representing worst performances. Scores for the total test is provided as a percentage of total points i.e. 108. In addition, 6 sub-systems scores can be generated separately in percentage of total score each representing a specific balance system
Spatiotemporal gait parameters | 6th week
  By using a stopwatch and measuring tape

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (2):
- Pakistan (2):
  - PhysioFit, Faisalabad, Punjab Province
  - Allied Hospital Faisalabad., Faisalābad, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersen EA, Stauss TG, Scowcroft JA, Brooks ES, White JL, Sills SM, Amirdelfan K, Guirguis MN, Xu J, Yu C, Nairizi A, Patterson DG, Tsoulfas KC, Creamer MJ, Galan V, Bundschu RH, Paul CA, Mehta ND, Choi H, Sayed D, Lad SP, DiBenedetto DJ, Sethi KA, Goree JH, Bennett MT, Harrison NJ, Israel AF, Chang P, Wu PW, Gekht G, Argoff CE, Nasr CE, Taylor RS, Subbaroyan J, Gliner BE, Caraway DL, Mekhail NA. Effect of High-frequency (10-kHz) Spinal Cord Stimulation in Patients With Painful Diabetic Neuropathy: A Randomized Clinical Trial. JAMA Neurol. 2021 Jun 1;78(6):687-698. doi: 10.1001/jamaneurol.2021.0538. PMID 33818600
- [Background] Castelli G, Desai KM, Cantone RE. Peripheral Neuropathy: Evaluation and Differential Diagnosis. Am Fam Physician. 2020 Dec 15;102(12):732-739. PMID 33320513
- [Background] Ferreira JSSP, Cruvinel Junior RH, Silva EQ, Verissimo JL, Monteiro RL, Pereira DS, Suda EY, Sartor CD, Sacco ICN. Study protocol for a randomized controlled trial on the effect of the Diabetic Foot Guidance System (SOPeD) for the prevention and treatment of foot musculoskeletal dysfunctions in people with diabetic neuropathy: the FOotCAre (FOCA) trial I. Trials. 2020 Jan 13;21(1):73. doi: 10.1186/s13063-019-4017-9. PMID 31931855
- [Background] Monteiro RL, Ferreira JSSP, Silva EQ, Donini A, Cruvinel-Junior RH, Verissimo JL, Bus SA, Sacco ICN. Feasibility and Preliminary Efficacy of a Foot-Ankle Exercise Program Aiming to Improve Foot-Ankle Functionality and Gait Biomechanics in People with Diabetic Neuropathy: A Randomized Controlled Trial. Sensors (Basel). 2020 Sep 9;20(18):5129. doi: 10.3390/s20185129. PMID 32916792
- [Background] Peterson M, Pingel R, Rolandsson O, Dahlin LB. Vibrotactile perception on the sole of the foot in an older group of people with normal glucose tolerance and type 2 diabetes. SAGE Open Med. 2020 Jun 13;8:2050312120931640. doi: 10.1177/2050312120931640. eCollection 2020. PMID 32587694
- [Background] Thukral N, Kaur J, Malik M. A Systematic Review and Meta-analysis on Efficacy of Exercise on Posture and Balance in Patients Suffering from Diabetic Neuropathy. Curr Diabetes Rev. 2021;17(3):332-344. doi: 10.2174/1573399816666200703190437. PMID 32619175
- [Background] Khan KS, Andersen H. The Impact of Diabetic Neuropathy on Activities of Daily Living, Postural Balance and Risk of Falls - A Systematic Review. J Diabetes Sci Technol. 2022 Mar;16(2):289-294. doi: 10.1177/1932296821997921. Epub 2021 Mar 14. PMID 33719603
- [Background] Akbari NJ, Naimi SS. The effect of exercise therapy on balance in patients with diabetic peripheral neuropathy: a systematic review. J Diabetes Metab Disord. 2022 Jul 4;21(2):1861-1871. doi: 10.1007/s40200-022-01077-1. eCollection 2022 Dec. PMID 36404857
- [Background] Prokai J, Murlasits Z, Banhidi M, Csoka L, Greci V, Atlasz T, Vaczi M. The Effects of a 12-Week-Long Sand Exercise Training Program on Neuromechanical and Functional Parameters in Type II Diabetic Patients with Neuropathy. Int J Environ Res Public Health. 2023 Apr 5;20(7):5413. doi: 10.3390/ijerph20075413. PMID 37048025
- [Background] Kang GE, Stout A, Waldon K, Kang S, Killeen AL, Crisologo PA, Siah M, Jupiter D, Najafi B, Vaziri A, Lavery LA. Digital Biomarkers of Gait and Balance in Diabetic Foot, Measurable by Wearable Inertial Measurement Units: A Mini Review. Sensors (Basel). 2022 Nov 29;22(23):9278. doi: 10.3390/s22239278. PMID 36501981